CLINICAL TRIAL: NCT00108238
Title: Estrogen Alternatives and Vascular Function in Post-Menopausal Women
Brief Title: Estrogen Alternatives Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CLIN-001-02F
Record Dates: First submitted 2005-04-14; First posted 2005-04-15 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2007-04

CONDITIONS: Healthy
Keywords: endothelial function; hormone replacement therapy; coronary flow reserve; posmenopausal women; women's cardiovascular heatlh
MeSH Terms: interventions — Raloxifene Hydrochloride

INTERVENTIONS:
Drug: Estradiol followed by progesterone
Drug: Raloxifene

SUMMARY:
Healthy postmenopausal women not currently taking hormone replacement or hormone modulating therapy take a 3-month course of estradiol/raloxifene/placebo to evaluate the effects of each on vascular function, as indicated by PET coronary flow reserve studies and brachial artery ultrasound, before and after use of the therapies. This is a randomized, placebo-controlled, blinded study.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women (no menses for greater than or equal to 12 months, or s/p [status post] hysterectomy with bilateral ovariectomy) not currently taking hormone replacement therapy (within previous 3 months)
* Normal mammogram within previous 12 months

Exclusion Criteria:

* Current or recent (within previous 3 months) hormone replacement therapy
* Current or recent (within previous 3 months) use of hormone alternatives such as raloxifene, tamoxifen, or soy estrogen preparations.
* LDL Cholesterol > 160 mg/dl.
* History of hypertension, diabetes mellitus, peripheral vascular disease, cerebrovascular disease, current smoking, history of DVT (deep vein thrombosis) or PE (pulmonary embolism), active gallbladder disease, family history of premature (men under 55 yrs, women under 65 yrs) coronary artery disease
* History of breast, uterine, or ovarian cancer Contraindication to adenosine administration (i.e., significant bronchospastic pulmonary disease, higher degree heart block)
* Inability to give informed consent
* Inability to temporarily (for 24 hours) discontinue potential vasoactive drugs, such as anti-inflammatory agents and aspirin, at least 24 hours prior to the examinations.
* History of coronary heart disease

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Dates: Start 2003-04; Study Completion 2006-12

CONTACTS AND LOCATIONS:
Overall Officials: Claire Duvernoy, M.D., Principal Investigator
Locations (1):
- VA Ann Arbor Healthcare System, Ann Arbor, Michigan, United States